CLINICAL TRIAL: NCT01278550
Title: Prevention of Recurrent Ulcer Bleeding in High-risk Users of Low-dose Aspirin (NSAID#2NANC Study)
Brief Title: Prevention of Recurrent Ulcer Bleeding in High-risk Users of Low-dose Aspirin
Status: Completed | Type: Observational
Sponsor: Chinese University of Hong Kong (Other)
Responsible Party: Principal Investigator, Francis KL Chan, professor, Chinese University of Hong Kong
Other Study IDs: 2NANC
Record Dates: First submitted 2011-01-18; First posted 2011-01-19 (Estimated); Last update posted 2015-08-13 (Estimated); Status verified 2015-08

CONDITIONS: Ulcer Hemorrhage

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No

GROUPS / COHORTS (2):
- Average risk cohort: Patients having no history of endoscopically confirmed ulcer bleeding, need long-term aspirin for cardiovascular or cerebrovascular prophylaxis and have H. pylori positive OR negative
- High risk cohort: Patients have history of endoscopically confirmed ulcer bleeding, need long-term aspirin for cardiovascular or cerebrovascular prophylaxis and have successful eradication of H. pylori based on histology

SUMMARY:
Low-dose aspirin is the mainstay of treatment for patients with coronary heart disease and stroke. However, low-dose aspirin increases the risk of ulcer bleeding. Current evidence indicates that 80 - 100 mg of aspirin daily provides good protection against vascular events and the risk of ulcer bleeding is low (about 1% per year). Since the overall risk of bleeding is low, aspirin users who do not have previous ulcer disease do not require prophylaxis with anti-ulcer drugs. In contrast, aspirin users with a history of ulcer disease have a 2- to 4-fold increased risk of ulcer bleeding. The best strategy for reducing the risk of bleeding in high-risk aspirin users remains unclear. Current strategies for high-risk patients include the use of anti-ulcer drugs, elimination of risk factors (e.g. Helicobacter pylori). Recently the investigators have shown that among aspirin users who are infected with H. pylori, the eradication of H. pylori is comparable to omeprazole, a proton pump inhibitor (PPI), in preventing recurrent ulcer bleeding in 6 months.

The investigators postulated that among patients with H. pylori infection and a history of ulcer bleeding who continue to use low-dose aspirin, the long-term risk of ulcer complications after eradication of H. pylori is comparable to that of average-risk aspirin users.

DETAILED DESCRIPTION:
Low-dose aspirin is increasingly used for the prophylaxis against coronary heart disease and stroke. However, it is also an important cause of peptic ulcer bleeding worldwide. In England and Wales, low-dose aspirin is estimated to account for about 10% of ulcer bleeding in people aged 60 and over [Weil 1995]. The problem of aspirin-related ulcer disease is expanding with the increasing use of aspirin for cardiovascular prophylaxis.

No dose of aspirin is entirely free of risk. Using a daily dose of aspirin as low as 75 mg, the risk of ulcer bleeding doubles that of non-users [Weil 1995]. Previous ulcer disease and concurrent major medical illnesses are important risk factors for ulcer bleeding with low-dose aspirin. Among aspirin users, those with previous ulcer disease have a 5-fold increased risk of ulcer bleeding [Lanas 2000]. Recently the investigators have shown that among aspirin users who are infected with H. pylori, the eradication of H. pylori is comparable to omeprazole in preventing recurrent ulcer bleeding in 6 months [Chan 2001]. However, whether curing H. pylori infection would confer long-term protection against ulcer bleeding for patients requiring life-long aspirin is uncertain.

To compare the long-term risk of ulcer complications in high-risk aspirin users after eradication of H. pylori with that of average-risk aspirin users. The latter is defined as patients who have no prior history of ulcer bleeding.

The investigators postulated that among patients with H. pylori infection and a history of ulcer bleeding who continue to use low-dose aspirin, the long-term risk of ulcer complications after eradication of H. pylori is comparable to that of average-risk aspirin users.

References Weil J, Colin-Jones D, Langman M, et al. Prophylactic aspirin and risk of peptic ulcer bleeding. Br Med J 1005;310:827-30.

Lanas A, Bajador E, Serrano P, et al. Nitrovasodilators, low-dose aspirin, other nonsteroidal antiinflammatory drugs, and the risk of upper gastrointestinal bleeding. N Engl J Med 2000;343:834-9.

Chan FKL, Chung SCS, Suen BY, et al. Preventing recurrent upper gastrointestinal bleeding in patients with Helicobacter pylori infection who are taking low-dose aspirin or naproxen. N Engl J Med 2001;344:967-73.

ELIGIBILITY:
High-risk cohort

Inclusion criteria:

Patients must fulfill ALL of the following:

1. History of endoscopically confirmed ulcer bleeding
2. Need long-term aspirin for cardiovascular or cerebrovascular prophylaxis
3. Successful eradication of H. pylori based on histology

Exclusion criteria:

1. Concomitant use of anti-ulcer drug, anticoagulant, non-aspirin NSAIDs or steroids
2. Previous acid-reduction gastric surgery
3. Gastric outlet obstruction, erosive esophagitis, gastroesophageal varices
4. Moribund or incurable cancers

Average-risk cohort

Inclusion criteria:

Patients must fulfill ALL of the following:

1. No history of ulcer bleeding
2. Need long-term aspirin for cardiovascular or cerebrovascular prophylaxis
3. H. pylori positive OR negative

Exclusion criteria:

1. Concomitant use of anti-ulcer drug, anticoagulant, non-aspirin NSAIDs or steroid
2. Previous acid-reduction gastric surgery
3. Moribund or incurable cancers
4. Previous attempts of H. pylori eradication

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: High-risk patients were from our hospital while average-risk patients were from our out-patient clinics
Sampling Method: Non-Probability Sample
Enrollment: 503 (Actual)
Dates: Start 1995-01; Primary Completion 2013-03 (Actual); Study Completion 2013-03 (Actual)

PRIMARY OUTCOMES:
Ulcer complications, defined as bleeding or perforation | 10 years

CONTACTS AND LOCATIONS:
Overall Officials: Francis KL CHAN, MD, Principal Investigator — Chinese University of Hong Kong
Locations (1):
- Prince of Wales Hospital, Hong Kong (sar), China